CLINICAL TRIAL: NCT01406067
Title: Treatment of Children With Peer Related Aggressive Behavior With the Treatment Programme THAV - a Randomized Controlled Trial
Brief Title: Treatment of Children With Peer Related Aggressive Behavior
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Manfred Doepfner, Manfred Doepfner, Prof. Dr., University of Cologne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: THAV-Study 1
Record Dates: First submitted 2011-07-26; First posted 2011-07-29 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Oppositional Defiant Disorder
Keywords: social skills training,; social competence training,; Oppositional Defiant Disorder; peer related aggressive behavior; randomized controlled trial
MeSH Terms: conditions — Oppositional Defiant Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Social Skills Training (Experimental)
  Interventions: Behavioral: Treatment Program for Children with Aggressive Behavior
- Play group (Active Comparator)
  Interventions: Behavioral: Play group

INTERVENTIONS:
Behavioral: Treatment Program for Children with Aggressive Behavior — 24 sessions with the child aiming at the reduction of peer related aggressive behavior via social skills training. Additionally up to 10 sessions with relatives of the child in most cases with the parents.
  Arms: Social Skills Training
Behavioral: Play group — 12 double sessions (totally 24 treatment hours) in groups with up to 5 children. Different play activities were presented including techniques to activate resources of the child. These interventions give the children the opportunity to train pro-social interactions. Additionally up to 3 parent sessions were also included.
  Arms: Play group

SUMMARY:
The efficacy of the Treatment Program for Children with Aggressive Behaviour (Therapieprogramm für Kinder mit aggressivem Verhalten, THAV) which is a social competence training delivered in an individual format will be evaluated in a randomized controlled trial with children aged 6 to 12 years with peer-related aggressive behaviour.

DETAILED DESCRIPTION:
The German Treatment Program for Children with Aggressive Behaviour (Therapieprogramm für Kinder mit aggressivem Verhalten, THAV) aims at the therapy of children aged 6 to 12 years with peer-related aggressive behaviour, which results in a persistent impairment of the relationships to other children. Contrary to other treatment approaches, this intervention aims at the individual treatment of problem maintaining and moderating factors of aggressive behaviour. Depending on the individual problem maintaining factors the treatment aims to modify social cognitive information processing, impulse control, social problem solving, social skills and social interactions. Methods: The efficacy will be tested in a partial randomized control group design with n=100 children. N=60 children will be treated for about half a year with the modules of THAV in weekly sessions. The control group of n=40 children will receive alternative interventions with group play and techniques to activate resources of the child. These interventions give the children the opportunity to train pro-social interactions. Outcome parameters are aggressive behaviour und comorbid symptoms as well as problem maintaining factors, psychosocial functioning, family burden and treatment satisfaction. Moreover, variables of the treatment process are assessed. Questionnaires, tests and individual problem checklist were used to assess these outcome and process parameters

ELIGIBILITY:
Inclusion Criteria:

* Age: 6 - 12 years
* IQ>= 80
* Diagnoses (ICD-10): F91, F92, F90.1
* high symptom score in the parent rated Symptom Checklist for Oppositional Defiant and Conduct Disorder (FBB-SSV) (Stanine ≥ 7) at assessment 1 and assessment 2
* Often conflicts with other children (clinical rating)
* Impaired social relationships / activities
* Parents agree in randomization
* in medicated children no planned change of the medication

Exclusion Criteria:

* other disorder is dominating
* other active psychotherapy
* severe mental disorder of the parents

Ages: 6 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change in Questionnaire for Aggressive Behavior of Children (FAVK) total score for peer related aggression | Change from pre- assessment to post assessment 30 weeks after treatment begin and to follow up 3 months and 9 months after post assessment
  The Questionnaire for Aggressive Behavior of Children (FAVK) is a newly developed parent rating scale which assesses several factors of peer related aggression: (1) disturbance of social cognitive information processing, (2) disturbance of social problem solving and social skills, (3) disturbance of impulse control, and (4) disturbance of social interaction. These scores a summed to a total score

SECONDARY OUTCOMES:
Change in Symptom Checklist for Oppositional Defiant and Conduct Disorder (FBB-SSV), parent and teacher rating | change form pre assessment to post assessment 30 weeks after treatment begin and follow up 3 months and 9 months after post assessment
  The Symptom Checklist for Oppositional Defiant and Conduct Disorder (FBB-SSV) assesses all symptom criteria for ODD and some of the symptom criteria of Conduct Disorders according to ICD-10 and DSM-IV.
Change in Child Behavior Checklist (CBCL) and Teacher Report Form (TRF) | change form pre assessment to post assessment 30 weeks after treatment begin and follow up 3 months and 9 months after post assessment
  The CBCL and the TRF are well evaluated rating scales for the assessement of a broad spectrum of child behavioral and emotional problems as perceived by parents and teachers respectively
Change in KINDL rating scale for quality of life | change form pre assessment to post assessment 30 weeks after treatment begin
  The KINDL is a German parent and patient rating scale for the assessment of different aspects of QoL
Change in Modified WFIRS (Weiss Functional Impairment Rating Scale) | change form pre assessment to post assessment 30 weeks after treatment begin
  The modified WFIRS is a parent rating scale for the assessment of psychosocial functioning in children with ODD/CD. The original WFIRS has been developed to assess psychosocial functioning in children with ADHD. Several items have been adapted or deleted in thise modified version.
Change in Individual Problem Checklist (IPC) | change form pre assessment to post assessment 30 weeks after treatment begin
  The IPC assesses individual problems as defined together with the parents. It represents the individual problems which were aimed to reduce with the treatment.
Change in Social Problem Solving Test (SPST) | change form pre assessment to post assessment 30 weeks after treatment begin
  The Social Problem Solving Test (SPST) is a newly developed test that assesses problem solving compentecies according to the social problem solving theory of Kenneth Dodge as well as behavioural tendencies in specific conflict situations.
Change in Five minutes speech sample (FMSS) | change form pre assessment to post assessment 30 weeks after treatment begin
  The FMSS is a standard assessment procedure to assess negative expressed emotions within the family. The parents are asked to describe their child for five minutes. The recorded descriptions were analyzed according to several domains.
Change in Depression Anxiety and Stress Questionnaire (DASS) | change form pre assessment to post assessment 30 weeks after treatment begin and follow up 3 months and 9 months after post assessment
  The DASS assesses parental depression anxiety and stress

CONTACTS AND LOCATIONS:
Overall Officials: Anja Goertz-Dorten, PhD, Principal Investigator — Department of Child and Adolescent Psychiatry Univ. Cologne
Locations (1):
- Department of Child and Adolescent Psychiatry at the University Cologne, Cologne, Germany

REFERENCES:
- [Derived] Katzmann J, Goertz-Dorten A, Hautmann C, Doepfner M. Social skills training and play group intervention for children with oppositional-defiant disorders/conduct disorder: Mediating mechanisms in a head-to-head comparison. Psychother Res. 2019 Aug;29(6):784-798. doi: 10.1080/10503307.2018.1425559. Epub 2018 Jan 19. PMID 29347904